CLINICAL TRIAL: NCT06950333
Title: The Development and Assessment of the Core Ultrasound Applications for Emergency Medical Technicians in Taiwan
Brief Title: Ultrasound Applications for Emergency Medical Technicians in Taiwan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202412164RINC
Record Dates: First submitted 2025-04-13; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Prehospital Emergency Medical Services; Point-of-care Ultrasound
Keywords: Prehospital ultrasound; emergency medical technicians; Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EMT who receive POCUS curriculum (Experimental): This arm includes certified advanced emergency medical technicians (EMT-P) who are enrolled in a structured point-of-care ultrasound (POCUS) education program developed specifically for prehospital providers in Taiwan. Participants receive a four-hour training module composed of didactic instruction and hands-on practice focused on trauma (FAST), dyspnea (lung ultrasound), suspected stroke (carotid Doppler), and cardiac arrest (focused cardiac ultrasound). Post-training assessments include written exams and objective structured clinical examinations (OSCEs). Participants will also complete follow-up assessments at six months and participate in supervised prehospital ultrasound scanning during real-world EMS missions.
  Interventions: Other: POCUS education curriculum

INTERVENTIONS:
Other: POCUS education curriculum — The training includes a 4-hour curriculum consisting of a 1-hour didactic session covering ultrasound principles and key applications, followed by 3 hours of hands-on practice using standardized models or phantoms under instructor supervision. Core scanning topics include Focused Assessment with Sonography for Trauma (FAST), lung ultrasound for dyspnea, carotid Doppler for suspected stroke, and focused cardiac ultrasound for cardiac arrest. Post-training assessments include a written test and an Objective Structured Clinical Examination (OSCE).

SUMMARY:
The goal of this prospective observational study is to develop and assess the core ultrasound applications for emergency medical technicians (EMTs) in Taiwan. The study focuses on advanced emergency medical technicians (EMT-Ps) and their ability to perform point-of-care ultrasound (POCUS) in prehospital settings.

The main questions it aims to answer are:

Can a standardized POCUS training program improve EMT-Ps' competency in ultrasound applications? What is the reliability and validity of the newly established POCUS assessment modules for EMT-Ps? Researchers will compare trained EMT-Ps' ultrasound proficiency and clinical decision-making before and after training to see if structured POCUS education enhances diagnostic accuracy and patient care in prehospital settings.

Participants will:

Attend a structured POCUS training program, including lectures and hands-on practice with standardized patients and simulation models.

Undergo competency assessments, including written exams, objective structured clinical examinations (OSCEs), and image interpretation tests.

Perform ultrasound scans on actual patients in prehospital settings, focusing on trauma, respiratory distress, stroke, and cardiac arrest cases.

Receive feedback and participate in follow-up assessments to evaluate knowledge retention and clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with one of the following conditions in the prehospital setting:

Trauma Dyspnea (shortness of breath) Suspected stroke Out-of-hospital cardiac arrest (OHCA)

Exclusion Criteria:

* Patients with hemodynamic instability or critical conditions requiring immediate resuscitation, making them unsuitable for focused prehospital ultrasound performed by EMT-Ps.
* Patients under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Image Quality Score for Target Structure Visualization | From enrollment to one day after patient was sent to hospital
  The score of ultrasound images assessing the visualization quality of target anatomical structures (e.g., blood vessels, Morrison's pouch, spleno-renal recess, cul-de-sac), evaluated using a standardized 10-point image quality rating scale (1 = Poor, 10 = Excellent). Each ultrasound image receives an overall score reflecting the adequacy of target structure visualization, as rated by trained reviewers.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nations JA, Browning RF. Battlefield applications for handheld ultrasound. Ultrasound Q. 2011 Sep;27(3):171-6. doi: 10.1097/RUQ.0b013e31822b7c14. PMID 21873854
- [Background] Brun PM, Chenaitia H, Gonzva J, Bessereau J, Bobbia X, Peyrol M; WINFOCUS (World Interactive Network Focused On Critical UltraSound) Group France. The value of prehospital echocardiography in shock management. Am J Emerg Med. 2013 Feb;31(2):442.e5-7. doi: 10.1016/j.ajem.2012.05.021. Epub 2012 Aug 4. No abstract available. PMID 22867834
- [Background] Fitzgibbon JB, Lovallo E, Escajeda J, Radomski MA, Martin-Gill C. Feasibility of Out-of-Hospital Cardiac Arrest Ultrasound by EMS Physicians. Prehosp Emerg Care. 2019 May-Jun;23(3):297-303. doi: 10.1080/10903127.2018.1518505. Epub 2018 Oct 17. PMID 30192687
- [Background] Mercer CB, Ball M, Cash RE, Rivard MK, Chrzan K, Panchal AR. Ultrasound Use in the Prehospital Setting for Trauma: A Systematic Review. Prehosp Emerg Care. 2021 Jul-Aug;25(4):566-582. doi: 10.1080/10903127.2020.1811815. Epub 2020 Sep 17. PMID 32815755